CLINICAL TRIAL: NCT02406898
Title: Operative Hysteroscopy for Fibroma by Classic Resection Versus Morcellation: a Ramdomised Study
Brief Title: Evaluation of a Hysteroscopic Morcellator in Hysteroscopic Treatment of Submucosal Fibroids
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-43
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-05

CONDITIONS: Evaluate Both Technics on Procedure Duration; Characteristics and Perioperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hysteroscopic surgery with morcellation technic (Experimental): The hysteroscope with the MH system will be introduced. Resection of fibroids or both will be realized. The procedure will end or when the fibroids will be completely resected.
  the procedure may be suspended before complete resection of fibroids or uterine perforation or higher operating time to 90 minutes or amount of liquid used distension than 9 liters or distension fluid deficit of more than one liter .
  Interventions: Device: morcellator uterine system (MH)Karl Storz, Tuttligen- Germany
- conventional hysteroscopy technic with resection. (Active Comparator): The hysteroscope with conventional resection system will be introduced. Resection of fibroids or both will be realized. The procedure will end or when the fibroids will be completely resected.
  the procedure may be suspended before complete resection of fibroids or uterine perforation or higher operating time to 90 minutes or amount of liquid used distension than 9 liters or distension fluid deficit of more than one liter (4 ).
  Interventions: Device: morcellator uterine system (MH)Karl Storz, Tuttligen- Germany

INTERVENTIONS:
Device: morcellator uterine system (MH)Karl Storz, Tuttligen- Germany

SUMMARY:
Hysteroscopic surgery is the gold standard for intra uterine pathology especially fibroma. Limit of this technic is duration of procedure which is correlated to operative complications. So, for patient with large fibrome or several fibromas, this technic is not indicated or performs in several times. A new technic of hysteroscopic surgery is available which is quicker than conventional technic. This technic is poorly evaluated. Aim of this study is to evaluate both technics on procedure duration.

DETAILED DESCRIPTION:
Material and Methods

We propose a monocentric-randomised study. Inclusion criteria are women over 18 years requiring hysteroscopic surgery for fibroma. After informed consent, patients will be randomised in two groups: hysteroscopic surgery with morcellation technic and conventional hysteroscopy technic with resection. The main objective is duration of procedure. Secondary objectives are characteristics and perioperative complications (distension media quantity, cervical injury, uterine perforation), immediate et long term postoperative data's (postoperative pain and synechia). We hypothesis hysteroscopic with morcellation reduces duration of procedure of 50%. The estimated size of population number is 30 per group and 60 for the study.

Expected results

We expected a significant decrease of procedure duration with hysteroscopic morcellation. This data will be interesting according peroperative complications are correlated to procedure duration and allow hysteroscopic surgery to patients with large or several fibromas.

ELIGIBILITY:
Inclusion Criteria:- Patient who is at least 18 years.

* Patient under effective contraception.
* Patient who underwent ultrasound confirming the presence of at least one or both uterine fibroids with a diameter less than 6 cm for the largest fibroid.
* Patient who underwent diagnostic hysteroscopy confirming the presence of one or two uterine fibroids classified as Type 0, 1 or 2 according to FIGO classification (10).
* Patient with an indication of intrauterine fibroid resection (bleeding disorders fetilité) by hysteroscopy.
* Patient who agreed to participate in the study and who signed informed consent.

Exclusion Criteria:

* Early Removal linked to patient's wish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
duration of procedure | intraoperative
  The duration of the operative hysteroscopy is the period between the first introduction and the last out of the hysteroscope.

SECONDARY OUTCOMES:
Distension fluid amount used during hysteroscopy | intraoperative
Cervical tear | intraoperative
The stopping rate of operative hysteroscopy before complete resection: | intraoperative
Postoperative pain upon awakening on a visual scale 0-10 | 6 hours after end of procedure
The postoperative adhesions rate diagnosed by hysteroscopy control | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Hôpital de la conception, Marseille, France